CLINICAL TRIAL: NCT04983290
Title: Clinical Trial to Assess the Effectiveness of the Food Plan Consisting of Products With Modified Consistency Called (Weancare-Domus) in Changing the Quality of Life in Patients With Parkinson's Disease
Brief Title: Outcomes to the Nutritional Need of Patients With Parkinson's Disease
Acronym: W-Domus
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Milko Zanini (Other)
Collaborators: Azienda Sanitaria Locale 3 Genovese (Other)
Responsible Party: Sponsor-Investigator, Milko Zanini, assistant professor, University of Genova
Organization: University of Genova (Other)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: W-DOMUS-PARK/2021
Record Dates: First submitted 2021-06-09; First posted 2021-07-30 (Actual); Last update posted 2021-09-28 (Actual); Status verified 2021-09

CONDITIONS: Deglutition Disorders; Parkinson Disease; Nursing; Quality of Life
MeSH Terms: conditions — Deglutition Disorders; Parkinson Disease

STUDY DESIGN:
Intervention Model Description: Randomized nutraceutical clinical trial controlled with cross-over design on two groups
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention (Experimental): The participating subjects belonging to the experimental group, will receive at home a set of foods with modified textures that allow the patient to feed for the observation period of 4 months, will also be followed by the dietary service of the center and by personnel identified within the protocol in order to verify compliance, liability and information regarding the evaluation scales involved in the project.
  Interventions: Dietary Supplement: weancare-domus
- control (No Intervention): The control group will continue with its own feeding for the entire observation period of the experimental group.

INTERVENTIONS:
Dietary Supplement: weancare-domus — Participants belonging to the experimental group will receive at home a set of foods that allows to receive the right amount of proteins and energy in a modified texture form to be prepared by themselves or by their caregivers
  Arms: intervention

SUMMARY:
The intervention involves the identification of 140 patients (70 per group), fed throughout the duration of the study with the two different solutions indicated. The subject will be interviewed by identified and trained personnel in order to collect the information and data required by the study with frequency indicated for the individual evaluation sheets. The subject himself will be provided with all the contact and availability information of the referents of the firm for the purpose of requesting information or reporting events. The subject in the studio will be contacted weekly in order to evaluate the trend by the study referents, according to his availability, and personally interviewed by staff belonging to the research group.

DETAILED DESCRIPTION:
Non-motor symptomatology in Parkinson's disease (PD) is related to the quality of life of patients . Malnutrition in the subject with Parkinson's is a still relevant variable that hesitates in sarcopenia and increased motor deficits in relation to loss of muscle mass and energy deficit. Guidelines from the European Society for Clinical Nutrition and Metabolism (ESPEN) recommend monitoring and implementing interventions in the presence of weight loss or body mass.

Disphagia is a syndrome common in Parkinson's patients, even in the early stages of the pathology. The study by Pflug and collaborators showed that only 5% of the patients observed were completely free from swallowing deficiency, while in 55% of subjects (66/119) aspiration or penetration of food and liquids in the airways were reported regardless of the stage of illness. Several studies, cited by Curtis and collaborators, show that the prevalence of disphagia varies between 11 and 97% of patients during the course of the disease. This condition affects both food safety, with the risk of aspiration and ab-ingestis, and malnutrition conditions, hydration deficiency, also affecting the overall survival of patients in relation to the onset of pneumonia.

From a nursing point of view, great interest has the integrated nutritional indices, easy and quick-to-use tools, which manage to determine promptly the presence and risk of malnutrition and which can be used daily in the patient's evaluation. The most suitable is the Mini Nutritional Assessment (MNA), which determines the risk of malnutrition before modification of biochemical parameters. MNA has a sensitivity of 96% and a specificity of 97%.

The adoption of scales that evaluate non-motorcycle-related symptoms helps to identify the sindromic dimension of the pathology, highlighting its components that impact the overall quality of life.

Patients who follow a level 3 and 4 modified texture diet of the IDDSI Framework scheme frequently encounter an overall reduction in energy and protein intake, determined by the way the meal is prepared in self-production, associated with an often drastic reduction in fluid intake with consequences in both systemic and specific terms for the gastrointestinal tract. Monitoring liquids introduced by subjects with swallowing deficiency is a Grade B recommendation in the ESPEN guidelines.

Disphagia is a frequent condition in the subject with Parkinson's disease, particularly in the advanced stages, recent studies begin to show a decay in the safety of swallowing and maintenance in the airway in these subjects, even in relatively early stages of the disease.

Therefore, the application of a specific nutritional program for patients with swallowing problems is recommended in the prevention of malnutrition in patients with Parkinson's disease. Previous studies showed the rapid reversibility of malnutrition in hospitalized elderly subjects with cognitive and functional impairment if enrolled in a specific nutritional program.

In view of the strong impact that eating difficulties have on the state of health of parkinson's disease patients suffering from disphagia, the widespread spread of dietary frailties related to the various degrees of disphagia and the importance that patients with slight difficulty swallowing or chewing do not develop further pathologies related to a nutritional deficit , it is necessary to study the effectiveness of specific nutritional programs developed to meet the person's need for nutrition The aim of the study is to improve the nursing-care management of Parkinson's disease patients with disphagia

ELIGIBILITY:
Inclusion Criteria:

* clinical diagnosis of FOIS-based disphagy or Smithard test (3 oz swallow test) (2 - 3) or previous FEES diagnosis
* classification of the functional oral intake scale (FOIS) level of disphagy in classes 4 or 5 (or levels 2-3 on specific clinical indication)
* Belonging to one of the territorial structures for the Management of Parkinson's Disease in the territory of Genoa

Exclusion Criteria:

* Terminally ill subjects for pathology
* Subjects with severe disphagia and indication to artificial nutrition (enteral/parenteral)
* Severe renal, liver and respiratory failure
* Disphagy level classifications inconsistent with inclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2021-11-01 (Estimated); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-05-30 (Estimated)

PRIMARY OUTCOMES:
Non-motor symptomatology change (Novel Non-Motor Symptoms Scale for Parkinson's Disease - NNMS) | 4 months
  Novel Non-Motor Symptoms Scale for Parkinson's Disease includes 9 domains and 30 items.
  Each symptom scored with respect to:
  Severity: 0 = None, 1 = Mild: symptoms present but causes little distress or disturbance to patient; 2 = Moderate: some distress or disturbance to patient; 3 = Severe: major source of distress or disturbance to patient.
  Frequency: 1 = Rarely (<1/wk); 2 = Often (1/wk); 3 = Frequent (several times per week); 4 = Very Frequent (daily or all the time).

SECONDARY OUTCOMES:
Suction and ab-ingestis events related to textured food change (Novel Non-Motor Symptoms Scale for Parkinson's Disease - Domain 6: Gastrointestinal tract) | 4 months
  Novel Non-Motor Symptoms Scale for Parkinson's Disease - Domain 6: Gastrointestinal tract includes 3 items.
  Each symptom scored with respect to:
  Severity: 0 = None, 1 = Mild: symptoms present but causes little distress or disturbance to patient; 2 = Moderate: some distress or disturbance to patient; 3 = Severe: major source of distress or disturbance to patient.
  Frequency: 1 = Rarely (<1/wk); 2 = Often (1/wk); 3 = Frequent (several times per week); 4 = Very Frequent (daily or all the time).
  19. Does the patient dribble saliva during the day? 20. Does the patient have difficulty swallowing? 21. Does the patient suffer from constipation? (Bowel action less than three times weekly)

OTHER OUTCOMES:
functional parameter related to malnutrition change: Gait speed | 4 months
  Gait speed in metres per second (m/s): the fastest gait speed in 4 metres after 3 trials was recorded. Patients may use an assistive device, if needed.
functional parameter related to malnutrition change: grip strength | 4 months
  grip strength of the hand in kg: Handgrip strength will assess using a hydraulic dynamometer. The participant will be seated, resting his or her arm on the chair arms and instructed to squeeze the dynamometer as hard as possible, with the highest score of the 3 trials recorded
functional parameter related to malnutrition change: muscle mass | 4 months
  muscle mass index (%) will be evaluate by Bioelectrical Impedance Analysis (BIA)
functional parameter related to malnutrition change: Body Mass Index (BMI) | 4 months
  weight in kg, height in cm (weight and height will be combined to report BMI in Kg/m^2)
functional parameter related to malnutrition change: arm circumference | 4 months
  arm circumference in cm
functional parameter related to malnutrition change: biomarkers | 4 months
  plasma cholinesterase concentration (U/ml)
functional parameter related to malnutrition change: biomarkers | 4 months
  plasma transferrin concentration (mg/dL)
functional parameter related to malnutrition change: biomarkers | 4 months
  plasma albumin concentration (g/dL)
functional parameter related to malnutrition change: immunological indices | 4 months
  lymphocyte count in 1 microliter (µL) of blood
functional parameter related to malnutrition change: Nutritional status evaluation | 4 months
  • phase angle and derived body composition data: Phase angle is a linear method of measuring the relationship between electric resistance (R) and reactance (Rc) in series or parallel circuits. It reflects cellular vitality and integrity, where normal values indicate preserved cellular activity. It is an important tool in assessing nutritional status in any situation, being superior to anthropometric and biochemical methods.
functional parameter related to malnutrition change: Nutritional status evaluation - MNA score | 4 months
  Mini Nutritional Assessment Score (MNA):Mini Nutritional Assessment score (MNA) is probably the most widely used and best validated score in different elderly populations and settings. The tool consists of a 6-item short form screening tool (MNA-SF) included in the 18-item long form scale (MNA-LF).
  From 24 to 30 points: Normal nutritional status; from 17 to 23.5 points: At risk of malnutrition; Less than 17 points: Malnourished
functional parameter related to malnutrition change: Bolus transit time evaluation | 4 months
  time of complete capture of the bolus and the reflex firing of swallowing in minutes

CONTACTS AND LOCATIONS:
Overall Officials: Marina Simonini, Dr, Principal Investigator — Asl 3 genovese
Locations (1):
- ASL 3 Genovese Struttura Complessa Recupero e Rieducazione Funzionale Ospedale "La Colletta" Via del Giappone, 5 - Arenzano (GE), Genova, Italy

IPD SHARING:
Plan to Share IPD: No